CLINICAL TRIAL: NCT05067257
Title: A Multicenter, Phase 2 Study to Assess the Safety and Efficacy of Epidural Resiniferatoxin for the Treatment of Intractable Pain Associated With Advanced Cancer
Brief Title: Study to Assess Epidural Resiniferatoxin for the Treatment of Intractable Pain Associated With Advanced Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sorrento Therapeutics filed for chapter 11 bankruptcy.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTX-CAP-201
Record Dates: First submitted 2021-09-17; First posted 2021-10-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pain, Intractable; Pain Cancer; Pain
Keywords: advanced cancer pain; cancer pain; pain; resiniferatoxin; RTX
MeSH Terms: conditions — Pain, Intractable; Cancer Pain; Pain | interventions — resiniferatoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Resiniferatoxin (Experimental): 15 mcg, 20 mcg, or 25 mcg in 2mL injected once into the epidural space
  Interventions: Drug: Resiniferatoxin
- Placebo (Placebo Comparator): 2mL injected once into the epidural space
  Interventions: Drug: Placebo
- Concurrent Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin is a compound purified from natural sources
  Other Names: RTX
  Arms: Resiniferatoxin
Drug: Placebo — Vehicle solution
  Arms: Placebo

SUMMARY:
This Phase 2 study assesses the safety and efficacy of a single injection of Resiniferatoxin versus placebo for the treatment of intractable advanced cancer pain.

DETAILED DESCRIPTION:
This is a global multicenter, randomized Phase 2 study for subjects with advanced cancer experiencing intractable pain to assess the safety and efficacy of a single epidural injection of Resiniferatoxin versus vehicle control. Additional subjects who elect to not enroll but are willing to be followed will comprise a Concurrent Control Group. Subjects will be followed for twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced cancer
* Targeted pain area of involvement that is at or below the lower thoracic or chest level down to lower extremities, attributed to the cancer
* If pain is present in other areas, able to differentiate pain in the target area is the primary source of pain
* Intractable pain that has not responded to standard therapies
* Be opioid tolerant, defined as an average daily opioid consumption > 30 mg oral morphine equivalent dose during the screening and which has been stable for the month prior to screening
* Have a Karnofsky Performance Scale score ≥ 50 at Screening
* In the Investigator's opinion, a reasonable expectation that the subject will be able to complete the study
* Able to comply with the study procedures and give informed consent
* Willing to follow contraception guidelines

Exclusion Criteria:

* Be undergoing or have plans to undergo changes to current cancer treatment from D-7 through M3
* Had an implantation of intrathecal pump or spinal cord stimulator less than 6 weeks prior to D1 or planning to undergo such a placement during the study prior to M3
* Have leptomeningeal metastases in the lumbar area
* Unless approachable via the caudal route, have the level of intended epidural injection within site of prior lumbar spine surgical procedures that could disrupt the epidural space or otherwise impair ability of the injection to reach nerves
* Has evidence of a non-correctable coagulopathy or hemostasis problem including a low platelet count, prothrombin time, abnormal PT or PTT, or on anticoagulant or antiplatelet therapies before and during investigational product (IP) administration
* Have evidence or history of bleeding disorder or disseminated intravascular coagulation, any recent hemorrhage or bleeding event within 4 weeks prior to D1
* Have abnormal neutrophil or serum creatinine
* Is febrile or has other evidence of infection within 24 hours of D1
* Has recently been diagnosed as COVID-19 positive or evidence of active infection. The subject may participate if full recovery has occurred with a negative RT-PCR test (any EUA cleared test) at least 1 week prior to D1
* Has an allergy or hypersensitivity to TRPV1 agonists, bupivacaine, radiographic contrast agents, fentanyl, hydromorphone, or morphine
* Pregnant at Screening or planning on becoming pregnant or currently breastfeeding
* Has an intrathecal shunt, increased intracranial pressure or evidence of brain pathology as determined by symptoms, history, physical examination, and/or magnetic resonance imaging (MRI)
* Is unable or distinguish the target pain from any additional loci of pain at screening
* Non-study related minor surgical procedure ≤ 2 days or major surgical procedure ≤ 7 days prior to screening and must be sufficiently recovered and stable prior to D1
* Has not recovered from toxicities from previous cancer treatment, including chemotherapy, hormone therapy, immunotherapy, radiotherapy or bisphosphonates. Participants are not eligible if they have received such therapy within the month prior to D1
* Non-study related minor surgical procedure ≤ 5 days or major surgical procedure ≤ 21 days prior to enrollment. In all cases, subjects must be sufficiently recovered and stable prior to IP administration on D1
* Arterial thrombi, myocardial infarction, admission for unstable angina, within 3 months prior to screening
* Clinically significant electrocardiogram abnormalities
* Have any medical condition that could adversely impact subject's participation or safety or interfere with pain assessments
* Participation in another investigational trial during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of any treatment-emergent adverse events of epidural Resiniferatoxin (RTX) [safety and tolerability] | Baseline through study completion at up to approximately 12 months
  To assess the safety of epidural RTX including incidence and severity of any short-term and long-term treatment-emergent adverse events (TEAEs) using the Common Terminology Criteria for Adverse Events (CTCAE) criteria

SECONDARY OUTCOMES:
Assess efficacy of RTX on pain associated with advanced cancer | Baseline through study completion at up to approximately 12 months
  To assess efficacy of each epidural RTX dose in comparison to control groups on the subject's intractable pain due to advanced cancer using the Brief Pain Inventory, Short Form (BPI-SF) score (1-10, with 10 associated with worse pain)
Assess RTX effect on quality of life | Baseline through study completion at up to approximately 12 months
  To assess the efficacy of each epidural RTX dose in comparison to control groups on the quality of life using Treatment Helpfulness Questionnaire score (graded 1-7, with 7 being most helpful)
Assess RTX effect on opioid consumption | Baseline through study completion at up to approximately 12 months
  To assess the effect of each epidural RTX dose on opioid consumption, measuring the average reduction compared to baseline of daily opioid consumption, calculated as an oral morphine equivalent dose

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (4):
- United States (4):
  - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - University of Florida, Gainesville, Florida
  - Oregon Health & Science University, Portland, Oregon
  - HD Research, Bellaire, Texas